CLINICAL TRIAL: NCT06291337
Title: Ibuprofen, a Phenylpropanoic Acid Nonsteroidal Anti-inflammatory Drug, Inhibits Human Sweet Taste and Glucose Detection
Brief Title: Ibuprofen Inhibits Human Sweet Taste
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rutgers, The State University of New Jersey (Other)
Collaborators: Monell Chemical Senses Center (Other)
Responsible Party: Principal Investigator, Paul A Breslin, Professor, Rutgers, The State University of New Jersey
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: Pro2019001483; 10-204Mc (Other: Rutgers IRB)
Record Dates: First submitted 2024-02-15; First posted 2024-03-04 (Actual); Last update posted 2024-03-04 (Actual); Status verified 2024-02

CONDITIONS: Treatment of Sweet Taste Receptors Without or With an Oral Rinse of Ibuprofen Solution in Healthy Participants; Treatment of Sweet Taste Receptors Without or With an Oral Rinse of Naproxen Solution in Healthy Participants

STUDY DESIGN:
Intervention Model Description: We are testing individual sin a within subject control for their sweet taste ratings of sugars without and with oral rinses of ibuprofen and naproxen.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment of sweet taste receptors with Ibuprofen oral rinse (Experimental): Participants were tested for sweetness perception without and with an oral rinse of ibuprofen.
  Interventions: Drug: Inhibition of Sweet Taste by Ibuprofen Oral Rinses
- Treatment of sweet taste receptors with naproxen oral rinse (Experimental): Participants were tested for sweetness perception without and with an oral rinse of naproxen.
  Interventions: Drug: Inhibition of Sweet Taste by Naproxen Oral Rinses

INTERVENTIONS:
Drug: Inhibition of Sweet Taste by Ibuprofen Oral Rinses — Participants rinse the mouth with ibuprofen and the impact on perceived sweet taste elicited by sugar solutions in the mouth was assessed
  Arms: Treatment of sweet taste receptors with Ibuprofen oral rinse
Drug: Inhibition of Sweet Taste by Naproxen Oral Rinses — Participants rinse the mouth with naproxen and the impact on perceived sweet taste elicited by sugar solutions in the mouth was assessed
  Arms: Treatment of sweet taste receptors with naproxen oral rinse

SUMMARY:
The sweet taste receptor, TAS1R2-TAS1R3, is expressed both orally, where it signals sweet taste, and extraorally in the intestine and pancreas, where it may affect glucose absorption and metabolism. Recently, ibuprofen and naproxen have been identified to inhibit human T1R3 when heterologously expressed in cells. In the present study, the initial objective was to determine if ibuprofen and naproxen inhibit interactions of sugars with human sweet taste receptor under normal, physiological conditions. Ten healthy participants were asked to rate sweetness intensity for a range of sweet stimuli (sucrose, fructose, sucralose) after a prerinse of ibuprofen, naproxen or water. Both ibuprofen and naproxen inhibited sweet taste intensity in a dose-dependent manner. In association studies, ibuprofen use has been linked to preserved metabolic function, as its use is correlated with lower rates of Alzheimer's disease, diabetes and colon cancer. Here the investigators present a potential novel pathway for systemic ibuprofen to impact these metabolic diseases.

DETAILED DESCRIPTION:
The sweet taste receptor, TAS1R2-TAS1R3, is expressed both orally, where it signals sweet taste, and extraorally in the intestine and pancreas, where it may affect glucose absorption and metabolism. Lactisole is a well characterized negative allosteric modulator of the transmembrane domain of T1R3. Lactisole binds with a phenylpropionic acid moiety. More recently, ibuprofen and naproxen, which are similar to lactisole in structure, have been identified to inhibit human T1R3 when heterologously expressed in cells. In the present study, the initial objective was to determine if ibuprofen and naproxen inhibit interactions of sugars with human sweet taste receptor under normal, physiological conditions. Ten healthy participants were asked to rate sweetness intensity for a range of sweet stimuli (sucrose, fructose, sucralose) after a prerinse of ibuprofen, naproxen or water. Both ibuprofen and naproxen inhibited sweet taste intensity in a dose-dependent manner. The experiment was repeated in vitro with TAS1R2-TAS1R3 expressing human cells, with ibuprofen reducing signaling of sucrose and sucralose. To explore ibuprofen's potential connection with glucose signaling and metabolism, the investigators next tested whether prerinses of lower concentrations of ibuprofen including a typical peak plasma concentrations (0.18 mM, 0.57 mM and 5.7 mM), would affect sweet taste intensity ratings of lower levels of glucose. Ibuprofen inhibited glucose sweetness in a dose dependent manner. Finally, the investigators tested whether prerinses of 0.12 mM and 0.24 mM ibuprofen (resulting from ingestion of two or three 200 mg pills respectively) affects detection thresholds of glucose, which are concentrations nearing post-prandial plasma glucose levels. Detection thresholds were significantly higher after rinsing with 0.24 mM ibuprofen compared to water rinses (p<0.01, n=12). In association studies, ibuprofen use has been linked to preserved metabolic function, as its use is correlated with lower rates of Alzheimer's disease, diabetes and colon cancer. Here the investigators present a potential novel pathway for systemic ibuprofen to impact these metabolic diseases.

ELIGIBILITY:
Inclusion Criteria:

* Participant must be able to taste sugars as sweet
* Participant must be able to make ratings on a scale and follow instructions

Exclusion Criteria:

* Participant must not be on any medications that would preclude exposure to NSAIDS
* Participant must not be on any medications that are know to alter taste perception

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2020-06-01 (Actual); Primary Completion 2023-09-01 (Actual); Study Completion 2023-09-30 (Actual)

PRIMARY OUTCOMES:
Sweet taste ratings | 6 months
  The impact of oral rinses with NSAIDS on sweet taste ratings of sugars on a labeled magnitude scale was assessed. The numeric outcome is the value of sweetness intensity provided by the participant from the labeled magnitude scale with each sweetener oral rinse.
Sugar detection thresholds | 6 months
  The impact of oral rinses with NSAIDS on detection thresholds for sugars was assessed. The detection threshold is the lowest concentration of the sweetener solution that can be distinguished from water. The numeric outcome is the concentration of sweetener solution that can be distinguished from water.

CONTACTS AND LOCATIONS:
Overall Officials: Paul A Breslin, Ph.D., Principal Investigator — Rutgers University
Locations (1):
- Food Science and Nutritional Sciences, New Brunswick, New Jersey, United States

IPD SHARING:
Plan to Share IPD: Yes
All of the individual participant data collected during the trial, after de-identification.
Supporting Information: Study Protocol
Time Frame: Immediately following publication and ending 7 years following article publication.
Access Criteria: Researchers who provide a methodologically sound proposal. Proposals should be directed to breslin@monell.org to request data to achieve aims of the proposal. Data are available for 7 years at a third party website:
URL: https://sites.rutgers.edu/breslin-lab/